CLINICAL TRIAL: NCT01745627
Title: 755nm Alex Laser for Treatment of Pigmented and Vascular Lesions and Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN11-PICO_RG2_PL
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Benign Pigmented and Vascular Lesions and Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser Treatment (Experimental)
  Interventions: Device: 755nm Alex laser

INTERVENTIONS:
Device: 755nm Alex laser

SUMMARY:
Evaluation of the safety and efficacy of the 755nm Alex laser for the treatment of benign pigmented and vascular lesions and scars

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between 18 and 85 years of age.
2. Subjects with Fitzpatrick skin types I to VI.
3. Subjects who have unwanted pigmented lesions, vascular lesions, striae and/or hypertrophic or atrophic scars
4. Subject who are willing to consent to participate in the study.

4.2 Exclusion Criteria

1. Subject who will not be photographed or who will not cooperate with the post treatment care and follow up schedule
2. Hypersensitive to light exposure.
3. Active localized or systemic infections.
4. Taking medication for which sunlight is a contraindication.
5. History of squamous cell carcinoma or melanoma.
6. History of keloid scarring.
7. Use of oral isotretinoin (Accutane®) within 12 months of initial treatment or during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment.
8. Prior treatment with laser or other devices in treatment area within 3 months
9. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
10. Subjects who are pregnant, have been pregnant within the last 3 months, are currently breast feeding or are planning a pregnancy within the study period.
11. Subjects that the physician determines ineligible based on standard of care treatment.

    -

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject ID was never assigned, so the # of subjects who started the subject was actually 1 less than what the protocol said.
Groups:
- Laser Treatment: 755nm Alex laser
Period: Overall Study
Arm/Group | Laser Treatment
Started | 42
Completed | 20
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Laser Treatment
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 24
  Race/Ethnicity: Asian | 6
  Race/Ethnicity: Hispanic | 9
  Race/Ethnicity: African American | 2
  Race/Ethnicity: Hispanic/Other | 1
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 4
    Fitzpatrick Skin Type II | 14
    Fitzpatrick Skin Type III | 14
    Fitzpatrick Skin Type IV | 6
    Fitzpatrick Skin Type V | 3
    Fitzpatrick Skin Type VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Clearance Based on Photographic Scale
Description: This scale ranges from 0 to 3, where 0 is 0-25% clearance, 1 is 26-50% clearance, 2 is 51-75% clearance and 3 is 76-100% clearance. The baseline picture was compared to a photograph taken at the follow up visit. The number of patients that fell into each category was recorded.
Time Frame: 1 months post last treatment
Population: 19 subjects were lost to follow up after their treatment. 2 subjects did not have clearance data but had photographs for each of the follow up visits. 4 subjects did not attend the 1 month follow up, but attended a 3 month follow up, so their data was included. 2 subjects were not included in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Laser Treatment
Number analyzed (Participants) | 15
Participants
  >75% | 2
  51-74% | 2
  26-50% | 4
  0-25% | 7

2. Primary Outcome: Clearance Based on Photographic Scale
Description: as for outcome 1
Time Frame: 3 months post last treatment
Population: 19 subjects were lost to follow up, 2 subjects did not have clearance data but had photographs for each of the follow up visits. 6 subjects did not have data for this follow up visit but had data for the 1 month follow up visit, so their data were included. 2 subjects were not included in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Laser Treatment
Number analyzed (Participants) | 13
Participants
  >75% | 2
  51-74% | 2
  26-50% | 4
  0-25% | 5

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured and followed for each patient's participation in the study, approximately 26 months.
Arm/Group | Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 17/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatment (N=42)
Redness (Skin and subcutaneous tissue disorders) | 5
Swelling (Skin and subcutaneous tissue disorders) | 1
Crusting (Skin and subcutaneous tissue disorders) | 6
Blistering (Skin and subcutaneous tissue disorders) | 6
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Puritis (Skin and subcutaneous tissue disorders) | 1
Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.